CLINICAL TRIAL: NCT06439290
Title: Voice Outcome of Glottoplasty, Cricothyroid Approximation, Thyroplasty, and Chondrolaryngoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ONZ-2024-0049/ONZ-2024-0081
Record Dates: First submitted 2024-05-14; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Surgery; Larynx; Transgenderism; Gender Dysphoria
Keywords: Transgender; Phonosurgery; Determinants; MRI
MeSH Terms: conditions — Laryngeal Diseases; Transsexualism; Gender Dysphoria | interventions — Laryngoplasty; Mastectomy

STUDY DESIGN:
Intervention Model Description: Purpose 1: prospective non-randomized controlled trial. Experimental group: persons undergoing phonosurgery Control group: age-matched PFAB/PMAB undergoing mastectomy/breast augmentation
  Purpose 2: Predictors of the outcome of abovementioned surgery in the experimental group will be determined using correlational research (regression analysis).
  Purpose 3: After optimization of MRI sequences and testing in healthy participants (n=5), a segmentation and measurement workflow will be completed. Objective measurement of pre- and postoperative laryngeal anatomy: Anatomical outcome measures will be obtained and compared before and one month/6 months after surgery in the experimental group.
Who Masked: Care Provider
Masking Description: Assessments will be performed by an ENT specialist and SLP of the research group who is blinded to study evolution and group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: phonosurgery (Experimental): Group undergoing phonosurgery (glottoplasty, cricothyroid approximation, thyroplasty or chondrolaryngoplasty)
  Interventions: Procedure: Phonosurgery
- Control group: other surgery (Active Comparator): Control group: age matched TGD PFAB/PMAB undergoing mastectomy or breast augmentation surgery with the same in- and exclusion criteria.
  Interventions: Procedure: Mastectomy/breast augmentation

INTERVENTIONS:
Procedure: Phonosurgery — Gender-affirming voice surgery (such as glottoplasty, cricothyroid approximation, thyroplasty and chondrolaryngoplasty), in addition to gender-affirming voice training and hormone therapy, plays an important role in achieving a gender-congruent voice in transgender and gender diverse people. In addition, these interventions are sometimes performed on cisgender men or women who wish to change their voice. However, the impact of these interventions on broad voice characteristics needs to be further investigated.
  Other Names: glottoplasty; thyroplasty; cricothyroid approximation; chondrolaryngoplasty
  Arms: Experimental group: phonosurgery
Procedure: Mastectomy/breast augmentation — Control group of PFAB and PMAB persons undergoing a mastectomy or breast augmentation surgery.
  Arms: Control group: other surgery

SUMMARY:
The purpose of this study is to measure the short- and long-term voice outcome and outcome predictors of glottoplasty, cricothyroid approximation, thyroplasty, and chondrolaryngoplasty using a prospective non-randomized controlled trial and a multidimensional voice assessment protocol. Secondly, a laryngeal magnetic resonance imaging protocol will be developed to measure pre- and postoperative anatomical factors and compare them with the acoustic changes.

DETAILED DESCRIPTION:
Gender-affirming voice surgery (such as glottoplasty, cricothyroid approximation, thyroplasty and chondrolaryngoplasty), in addition to gender-affirming voice training and hormone therapy, plays an important role in achieving a gender-congruent voice in transgender and gender diverse people. In addition, these interventions are sometimes performed on cisgender men or women who wish to change their voice. However, the impact of these interventions on broad voice characteristics needs to be further investigated.

A thyroid chondroplasty is a procedure in which the cartilage of the larynx is flattened to make the larynx ("Adam's apple") less visible. This procedure is sometimes performed in combination with voice surgery. Although clinically in some cases we observe a temporary lowering of the pitch of the voice during thyroid chondroplasty, little is known in the literature about the impact of this surgery on voice characteristics.

The first purpose is to measure the effect of glottoplasty, cricothyroid approximation, thyroplasty and/or thyroid chondroplasty on a) acoustic voice characteristics (such as the pitch and resonance of the voice), b) perception of femininity/masculinity, c) psychosocial well-being and satisfaction and d) the function of the vocal folds.

Persons undergoing a glottoplasty, cricothyroid approximation, thyroplasty and/or thyroid chondroplasty in the head and neck surgery department are routinely invited to several pre- and postoperative check-up appointments in the head and neck surgery and ear, nose and throat department. These people will be invited to participate in the study in which the data, which are routinely collected preoperatively, 1 week, 1 month, 6 months and 12 months postoperatively during a speech-language pathology (SLP) consultation and a head and neck surgery consultation. These data will be used for scientific research to study the outcome of such surgery on phonation. These pre- and post-operative consultations are clinically standard. During these consultations, a voice assessment and videolaryngostroboscopic examination of the vocal folds are routinely performed.

Recordings and images obtained through these studies can be further processed in the context of this scientific research (such as conducting a listening experiment, analyzing (e.g. using the VALI form) and measuring the video laryngostroboscopy results, etc.).

Secondly, factors (determinants) that influence the effect of previous surgical interventions will be studied within this research.

The third purpose of this study is to develop and validate a laryngeal magnetic resonance imaging (MRI) protocol using a laryngeal surface coil to measure pre- and postoperative anatomical factors (vocal fold length and thickness, thyroarytenoid muscle mass and area) and compare them with the acoustic changes.

ELIGIBILITY:
PURPOSE 1:

Inclusion criteria for surgery participants:

* Persons who will soon undergo surgery on the vocal folds and/or larynx (including glottoplasty, cricothyroid approximation, thyroplasty and/or thyroid chondroplasty) at UZ Gent
* At least 18 years old
* Sufficient command of the Dutch language for understanding the informed consent letter and completing Dutch questionnaires

Inclusion criteria for volunteers to provide speech samples:

- Cisgender men or women

Inclusion criteria for volunteer listeners for the listening experiment:

* Dutch-speaking
* Self-reported normal hearing

PURPOSE 2: same as above.

PURPOSE 3:

Inclusion criteria for the healthy participants:

* At least 18 years old
* Sufficient command of the Dutch language to complete a Dutch questionnaire

Exclusion criteria for the healthy participants:

- One or more contraindications for an MRI examination. These contraindications are checked using a questionnaire (safety checklist).

Inclusion criteria for the pre- and postoperative MRI participants:

- Random selection of +- 10 participants of purpose 1.

Exclusion criteria for the pre- and postoperative MRI participants:

- One or more contraindications for an MRI examination. These contraindications are checked using a questionnaire (safety checklist).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons with both a masculine/feminine/nonbinary gender identity
Enrollment: 290 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Speaking fo | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Speaking fundamental frequency
FF 1-5 | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Formant frequencies 1-5
Perceptual femininity/masculinity score | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Self-perception and listener perceptions of femininity and masculinity. Visual analogue scale (0 = very masculine, 100 = very feminine).

SECONDARY OUTCOMES:
Vocal capacity | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Dysphonia Severity Index, cut-off score 1.6 (above 1.6 is normophonic)
Vocal range | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Voice Range Profile (min-max of fo and intensity (SPL))
Vocal quality | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Acoustic Voice Quality Index, cut-off score 2.95 (below 2.95 is normophonic)
Laryngeal function | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Flexible videolaryngostroboscopy
PROMs: Voice Handicap Index | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Voice Handicap Index, score from 0-120, the higher the score, the worse.
PROMs: Trans Woman Voice Questionnaire | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Trans Woman Voice Questionnaire, score from 1-120, the higher the score, the worse.
Other PROMs | pre, post 1 (1 week), post 2 (1 month), post 3 (6 months), post 4 (1 year)
  Visual analogue scales to measure satisfaction (VAS with 0=strongly disagree, 100=strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Clara Leyns, PhD, Study Director — University Ghent; Evelien D'haeseleer, PhD, Principal Investigator — University Ghent; Peter Tomassen, PhD, MD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent, East-Flanders
  - Ghent University, Ghent, East-Flanders

IPD SHARING:
Plan to Share IPD: No